CLINICAL TRIAL: NCT05869435
Title: A First-in-human, Single-arm, Single-center, Feasibility Study to Assess the Efficacy and Safety of the FastWire REvascularisation of Extremities, (For LOWer Limbs) (FREEFLOW)
Brief Title: FastWire REvascularisation of Extremities, (For LOWer Limbs) - Feasibility Study (FREEFLOW)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Versono Medical Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIP001FREEFLOW
Record Dates: First submitted 2023-05-11; First posted 2023-05-22 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Chronic Total Occlusion of Arteries of the Extremities
Keywords: Chronic Total Occlusion; Peripheral; CTO; FastWire System; FastWire Guidewire; intra-luminal; Active wire; Procedure; Device

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- FastWire System - Peripheral (Other): This study is to assess the safety and efficacy of the FastWire System. It is intended to assess that the FastWire System can facilitate the intra-luminal placement of conventional guidewires or treatment devices beyond peripheral artery chronic total occlusions (CTOs). This is a First in Human study
  Interventions: Device: FastWire System Device - Peripheral

INTERVENTIONS:
Device: FastWire System Device - Peripheral — The Investigator can use the FastWire System during the procedure to cross CTO Caps and/or to cross multiple lesions.

SUMMARY:
This study is to assess the safety and efficacy of the FastWire System. It is intended to assess that the FastWire System can facilitate the intra-luminal placement of conventional guidewires or treatment devices beyond peripheral artery chronic total occlusions (CTOs)

DETAILED DESCRIPTION:
A first-in-human, single-arm, single-center, feasibility study to assess the efficacy and safety of the FastWire System in patients who have a chronic total occlusion in their peripheral vasculature causing an ischemic limb. The enrollment will consist of up to 10 patients meeting the inclusion/exclusion criteria.

ELIGIBILITY:
Inclusion Criteria:

1. The patient, or the patient's legal guardian has signed and dated an Informed Consent Form.
2. Aged between 18 years and 85 years (inclusive).
3. Severe claudication assessed as Rutherford category 3 or CLTI assessed as Rutherford category 4 or 5 LEAD.
4. Angiographic confirmation of a de novo, CTO, infrainguinal ligament including above the knee, below the knee, or below the ankle vessels.

Exclusion Criteria:

1. Life expectancy of less than 12 months.
2. Females who are pregnant or lactating (urine test for women of childbearing age).
3. Myocardial infarction or stroke in two months prior to the index procedure.
4. Known, unstable coronary artery disease or other, uncontrolled comorbidity.
5. Any known haemorrhagic or coagulation deficiency.
6. Evidence of active infection, including but not limited to the target limb.
7. Current use of cocaine or other substance of abuse.
8. Patients who have received any thrombolytic therapy in the last two weeks.
9. History of severe allergy or contraindication, to contrast medium or other medications used during or after endovascular therapy.
10. Subject participating in another study involving an investigational drug or device
11. Patient has surgery or vascular intervention planned within 30 days of the index procedure.
12. Patient has had a previous peripheral bypass that includes the target vessel.
13. Patient has had a previous intervention in the target CTO (angioplasty, stenting) including at time of index procedure.
14. Patient tests positive for coronavirus disease (COVID-2019), as per site standard practice.
15. Estimated Glomerular Filtration Rate (eGFR) of less than 30 ml/min.
16. Platelet count < 50,000.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2022-12-14 (Actual); Primary Completion 2022-12-16 (Actual); Study Completion 2023-01-17 (Actual)

PRIMARY OUTCOMES:
Technical Success (On Procedure Day) | Day 1
  Ability of the FastWire to successfully cross angiographically confirmed chronic total occlusions and provide a platform for delivery of other treatment devices.
Clinical success (On Procedure Day) | Day 1
  Clinical success is assessed as the angiographically confirmed passage of the FastWire tip through the lesion and the successful delivery and retrieval of FastWire and the delivery of a treatment device to the target site.
Freedom from Serious Adverse Events related to the use of FastWire, at 30 days post procedure: | Up to Day 30
  * Cardiovascular deaths.
  * Vessel dissection requiring an intervention to resolve.
  * Unplanned index limb amputation.
  * Symptomatic distal embolization.

SECONDARY OUTCOMES:
Freedom from Serious Adverse Device Effects (SADE) (Up to Day 30) | Up to Day 30
  Freedom from Serious Adverse Device Effects (SADE).
Freedom from Vessel dissection or bleeding (Within 24 Hours) | Within 24 Hours
  Freedom from Vessel dissection or bleeding within 24 hours (16-36 hours) of index procedure.
Procedural success (On Procedure Day) | Day 1
  Procedural success, defined as achievement of technical success together with post procedure patency (less than 50% residual diameter stenosis of target vessel patent as assessed by angiographic imaging post device retrieval.
Procedure related mortality (Up to Day 7 & Day 30) | Up to Day 7 & Day 30
  All procedure related mortality at day 7 post procedure, and all-cause mortality at 30 days post procedure.

CONTACTS AND LOCATIONS:
Locations (1):
- INDEN, Santo Domingo, Dominican Republic

IPD SHARING:
Plan to Share IPD: No